CLINICAL TRIAL: NCT02586857
Title: A Phase 1b/2, Multicenter, Open-label Study of ACP-196 in Subjects With Recurrent Glioblastoma Multiforme (GBM)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-209
Record Dates: First submitted 2015-10-17; First posted 2015-10-27 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; GBM; Btk,; CLL; Chronic Lymphocytic Leukemia; NK; Natural Killer (Cells); ORR; Overall Response Rate; OS; Overall Survival; RANO; Response Assessment in Neuro-oncology (Criteria); RCI; Reliale Change Index (methodology)
MeSH Terms: conditions — Glioblastoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): ACP-196 200 mg administered orally (PO) twice per day (BID)
  Interventions: Drug: ACP-196
- Cohort 2 (Experimental): ACP-196 400mg administered orally (PO) once per day (QD).
  Interventions: Drug: ACP-196

INTERVENTIONS:
Drug: ACP-196 — Cohort 1: ACP-196 200 mg (PO) twice per day (BID) Cohort 2: ACP-196 400 mg (PO) once per day (QD).
  Other Names: Acalabrutinib.

SUMMARY:
A Phase 1b/2, Multicenter, Open-Label Study of ACP-196 in Subjects with Recurrent Glioblastoma Multiforme (GBM)

DETAILED DESCRIPTION:
A Phase 1b/2, multicenter, open-label study was designed to evaluate the efficacy and safety of acalabrutinib in subjects with recurrent glioblastoma multiforme (GBM) who had progressed after one or two prior systemic treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Histologically confirmed GBM at first or second recurrence after concurrent or adjuvant chemotherapy or radiotherapy (must have received temozolomide).
* Radiographic demonstration of disease progression by MRI following prior therapy.
* Measurable disease (bidimensional) as defined by the RANO criteria, with a minimum measurement of 1 cm in longest diameter on MRI performed within 21 days of first dose of acalabrutinib; MRI must have been obtained ≥4 weeks after any salvage surgery after first or second relapse.
* Stable or decreasing dose of corticosteroids ≥5 days before baseline MRI (at study entry).
* On a stable dose of any required therapy (such as anticonvulsant medication for subjects to be enrolled into the Phase 1b portion), for ≥3 weeks before the first dose of acalabrutinib.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Life expectancy ≥ 12 weeks.
* Completion of all prior anticancer therapy before first ACP-196 dose.
* Need to have recovered (i.e., Grade ≤1 or baseline) from AEs associated with prior cancer therapy. Note: Subjects with Grade ≤2 neuropathy or Grade

  * 2 alopecia are an exception, and may qualify for the study.

Exclusion Criteria:

* Three or more prior lines of systemic therapy for GBM.
* Prior malignancy (other than GBM), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥2 years. Any cases of prior malignancy allowed on study are to be approved by the study medical monitor.
* Significant cardiovascular disease.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Evidence of bleeding diathesis or coagulopathy.
* Requires urgent palliative intervention for primary disease
* Requires treatment with a strong CYP3A4 inhibitor..
* History of stroke or clinically significant intracranial hemorrhage within 6 months before first dose of study drug.
* Breastfeeding or pregnant.
* Subjects previously treated with bevacizumab (Avastin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (5):
- United States (5):
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-ST-209&attachmentIdentifier=eb0e1db1-4c84-4dd3-bbd8-1cb9943a1caf&fileName=ACE-ST-209_redactedCSP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Acalabrutinib: Acalabrutinib 200mg PO BID.
- Cohort 2 - Acalabrutinib: Acalabrutinib 400mg PO QD.
Period: Overall Study
Arm/Group | Cohort 1 - Acalabrutinib | Cohort 2 - Acalabrutinib
Started | 15 | 9
Enrolled | 15 | 9
Received Study Medication | 15 | 9
Discontinued Study | 14 | 9
Completed | 14 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Acalabrutinib 200mg administered orally (PO) twice daily (BID).
- Cohort 2: Acalabrutinib 400mg PO (QD).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: Year] | 58.7 (6.74) | 45.7 (13.84) | 53.8 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 7 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Tumor Status for Overall Response Rate With Use of RANO Criteria.
Description: To evaluate the efficacy of acalabrutinib monotherapy in subjects with recurrent GBM based on overall response rate (ORR) per the Response Assessment in Neuro-oncology (RANO) criteria. Responses are either complete response (CR) or partial response (PR) by RANO.
Time Frame: On Cycle 3 Day 1, Cycle 4 Day 1 (4 weeks after Cycle 3 Day 1 scan to evaluate for response stability), then on Day 1 of every other cycle (every 8 weeks) thereafter (e.g., Cycle 6 Day 1, Cycle 8 Day 1)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Acalabrutinib 200mg by PO BID.
- Cohort 2: Acalabrutinib 400mg by PO QD.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 15 | 9
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include starting on or after Day 0 and on or before Day 940.
Groups:
- Cohort 2 - Acalabrutinib: Acalabrutinib 400mg PO (QD)
Arm/Group | Cohort 1 | Cohort 2 - Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 12/15 | 7/9
Serious Adverse Events (participants affected / at risk) | 6/15 | 4/9
Other Adverse Events (participants affected / at risk) | 15/15 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=15) | Cohort 2 - Acalabrutinib (N=9)
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Influenze (Infections and infestations) | 0 | 1
Streptococcal (Infections and infestations) | 0 | 1
Abdominal Infection (Infections and infestations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=15) | Cohort 2 - Acalabrutinib (N=9)
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Vision Blurred (Eye disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Fatigue (General disorders) | 6 | 3 — General Disorders and Administration Site Conditions.
Catheter Site Pain (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions.
Gait Disturbance (General disorders) | 1 | 1 — General Disorders and Administration Site Conditions.
Mucosal Inflammation (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions.
Oedema Peripheral (General disorders) | 3 | 1 — General Disorders and Administration Site Conditions.
Chest Discomfort (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Chest Pain (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Feeling Cold (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Non-Cardiac Chest Pain (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions.
Hordeolum (Infections and infestations) | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Tinea Pedis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
CD4 Lymphocytes Decreased (Investigations) | 1 | 2
Platelet Count Decreased (Investigations) | 0 | 1
Vitamin D Decreased (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 1
Lymphocyte Count Decreased (Investigations) | 3 | 1
Alanine Aminotransferase Increased (Investigations) | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 7 | 5
Aphasia (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 2
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 4 | 0
Parosmia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Cognitive Disoder (Nervous system disorders) | 0 | 1
Disturbance in Attention (Nervous system disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Apiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Aceneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hot Flush (Vascular disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02586857/Prot_003.pdf
  • Statistical Analysis Plan (2018-04-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02586857/SAP_001.pdf